CLINICAL TRIAL: NCT00388687
Title: Hypoxia Imaging With the Novel Radiopharmaceutical 18F Fluoroazomycin Arabinoside (FAZA)- Prognostic Impact in Cervical Cancer
Brief Title: Hypoxia Imaging With 18F FAZA. Prognostic Impact in Cervical Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Medical University of Vienna (Other)
Other Study IDs: EK Nr: 241/2006
Record Dates: First submitted 2006-10-16; First posted 2006-10-17 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-10

CONDITIONS: Uterine Cervical Neoplasms
Keywords: Hypoxia; FAZA; PET; Radiochemotherapy
MeSH Terms: conditions — Uterine Cervical Neoplasms; Hypoxia | interventions — fluoroazomycin arabinoside

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Prospective

INTERVENTIONS:
Drug: 18F Fluoroazomycin Arabinoside (FAZA)

SUMMARY:
The aim of this study is to visualize the tumor hypoxic tissue, the potential quantitative changes and the biological behavior of cervical carcinoma (primary and / or lymph nodes) before, during and after radiochemotherapy with the novel hypoxia PET tracer 18FAZA.

DETAILED DESCRIPTION:
Introduction

Tumor hypoxia has been shown to be a prognostic factor for local progression and prognosis in several types of human cancers (1-4), including cervical carcinoma (5). Distribution of oxygen within a tumor can diminish toward the less vascularized center of the tumor (6, 7).

Hypoxia is an important factor in many pathological processes, including tumor formation, where it has been associated with resistance to radiotherapy, malignant progression, and metastasis. Although hypoxia is toxic to both cancer and normal cells, cancer cells undergo genetic and adaptive changes that allow them to survive and even proliferate within a hypoxic environment. These processes contribute to the malignant phenotype and to aggressive tumor behavior.

Hypoxia has a negative effect on anti cancer treatment (8). Radiotherapy is a major treatment modality for advanced cervical carcinomas and requires free radicals from oxygen to destroy target cells, and cells in hypoxic areas were found to be resistant to radiation-induced cell death (9). The gold standard for measuring hypoxia in tumors is the invasive technique of using computerized oxygen-sensitive electrodes. This method is cumbersome and expensive and has not become a general clinical tool for hypoxia measurement (10, 11).

Positron emission tomography (PET) becomes an interesting and promising diagnostic modality for hypoxia imaging in tumor tissue. Several tracers were developed for this purpose and Fluoromisonidazole (18FMISO) is the most extensively hypoxia tracer studied both in humans and animals (12-15). Previous results for imaging hypoxia using FMISO showed the regional distribution of tumor hypoxia, expressed as fractional hypoxic volume (16). However, its major disadvantages lie on its slow clearance kinetics and its high lipophilicity.

18Ffluoroazomycinarabinofuranoside (18FAZA) is recently synthesized and introduced as a hypoxia tracer in various tumor-bearing mice using PET and autoradiography with promising results. (17). 18FAZA showed also superior biokinetics in comparison to 18F-MISO in animals (18). The safety and feasibility of FAZA was evaluated recently in 10 patients with advanced squamous cell carcinoma of the head and neck. The authors of this study concluded that PET imaging with FAZA appears to be safe and feasible in patients with head and neck tumors. (19).

Aim of the study

The aim of this study is to visualize the tumor hypoxic tissue, the potential quantitative changes and the biological behavior of cervical carcinoma (primary and / or lymph nodes) before, during and after radiochemotherapy with the novel hypoxia PET tracer 18FAZA.

Materials and methods

Patients

Twenty-five patients with cervical carcinoma (T2Nx or TxN1) will be included in the present study. In addition to the routine pre-therapeutical staging of cervical cancer, 18FAZA PET will be performed before, during the planed radio/chemotherapy (short before brachytherapy) and 3 months after the therapy.

Synthesis and quality control 18FAZA (Research Center Seibersdorf)

18FMISO will be synthesized as previously described (20). The synthesis of 18F-FAZA will be performed as follows (21):5 mg of the precursor 1-(2,3-diacetyl-5-tosyl-a-D-arabinofuranosyl)-2-nitroimidazole in 1 mL of dimethyl sulfoxide were reacted with the mixture of azeotropically dried 18F-fluoride, 15 mg of Kryptofix 2.2.2. (Merck), and 3.5 mg of K2CO3 at 100C for 5 min. After hydrolysis with 1 mL of 0.1 N NaOH (2 min,30C), 0.5 mL of 0.4N NaH2PO4 was added for neutralization. The product was purified first using an alumina cartridge (Alu N light; Waters) and then high performance liquid chromatography (HPLC) (Phenomenex Nucleosil C18; ethanol/NaH2PO4 buffer (5:95); flow, 4mL/min; detection ultraviolet (320nm), Na(Tl)). The product was obtained in radiochemical yields of 20.7%+-3.5% (n=12) at end of the beam. After irradiations of 1 h at 35µA, 9.1 +-1.4GBq (n=8) 18FFAZA will be isolated.

[18F]FAZA PET imaging

Patients

18FFAZA imaging will be performed in all patients after overnight fasting on a dedicated full ring PET scanner (Advance, General Electric Medical Systems, Milwaukee, WI). The patients will be scanned subsequent to the administration of the activity (dynamic scan) and 2 hours afterwards (static scan). For each image acquisition a 10-min transmission scan will be performed. All images will be acquired in a 3D-mode with a matrix of 128x128. The dynamic scan (pelvis) begins with the intravenous administration of 370 MBq 18FFAZA. Over the first hour 21 frames will be acquired (6 frames 20s, 6 frames 30s, 2 frames 150s, 4 frames 300s, 3 frames 600s). Two hours after the application a 10-min static scan (pelvis + abdomen) will be acquired. The images are reconstructed using an iterative algorithm (OSEM). In addition to visual interpretation of the acquired images a semi quantitative analysis will be performed by drawing regions of interest (ROIs) in tumor tissue (primary and lymphnodes). For these ROIs both a standardized uptake value (SUV) and ratios to normal tissue (muscle) will be calculated.

Blood sampling

Simultaneously to the FAZA PET scans blood sampling (10ml) will be drawn for measurements of protein concentrations (VEGF, Osteopontin, PAI). In total, 30 ml blood will be collected from each patient.

Radiation burden

The estimated radiation burden for 18FFAZA (370MBq) examination amounts about 12 mSv (equivalent to a CT examination of the thorax).

Risks, Side effects, Toxicity

The fluorine-18(18F) labeled compound is obtained by nucleophilic substitution of a tosylate-precursor with no-carrier-added 18F-fluoride in a specific activity of > 74 MBq / nmol. The administration of 370 MBq 18F-FAZA will therefore correspond to < 5 nmol compound and will not exert any pharmacologic or toxicologic effect. Similar radiopharmaceutical such as 18FMISO showed no side effects in their clinical use in human (22)

Including criteria for patients

First diagnosis of histologically proven cervical cancer FIGO stage IB2 to IVA. Treatment intention for the purpose of achieving cure Age < 80 years No previous standard or radical hysterectomy

Excluding criteria for patients

Pregnancy, breast-feeding women, patients that are not able to lie motionless for one hour.

Palliative treatment, recurrent disease, neoadjuvant chemotherapy, other pre-existing malignancies, age > 80 years,

Statistics (SUVs)

Results will be given as median (range). The t-test will be used for comparison of groups, and a p value <0.05 is considered significant.

"Median SUV": stands for the median of the maximal SUVs of particular regions of interest (ROI).

ELIGIBILITY:
Inclusion Criteria:

* First diagnosis of histologically proven cervical cancer FIGO stage IB2 to IVA.
* Treatment intention for the purpose of achieving cure
* Age < 80 years
* No previous standard or radical hysterectomy

Exclusion Criteria:

* Pregnancy, breast-feeding women, patients that are not able to lie motionless for one hour.Palliative treatment, recurrent disease, neoadjuvant chemotherapy, other pre-existing malignancies, age > 80 years,

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25
Dates: Start 2006-07; Study Completion 2007-07

CONTACTS AND LOCATIONS:
Overall Officials: Georgios Karanikas, Prof. M.D., Study Director — Medical Universitiy of Vienna
Locations (2):
- Austria (2):
  - Medical Universitiy of Vienna, Vienna
  - Medical University of Vienna, Vienna